CLINICAL TRIAL: NCT01184131
Title: Implementation and Evaluation of Formal Training for Mentors of K-Series Mentored Career Awards
Brief Title: NCRR ARRA Development-Workforce Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: H-2009-0146; 3UL1RR025011-03S2 (NIH)
Record Dates: First submitted 2010-08-10; First posted 2010-08-18 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Research Mentoring Skills
Keywords: Mentor Training; Randomized trial of mentoring effectiveness; Mentoring clinical researchers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mentor Training (Experimental): The group that is randomized into the intervention group to attend Mentor Training Sessions.
  Interventions: Other: Mentor Training
- No Mentor Training (No Intervention)

INTERVENTIONS:
Other: Mentor Training — Four 2 hour sessions of Mentor Training
  Arms: Mentor Training

SUMMARY:
The research proposed in this collaborative application Implementation and Evaluation of Formal Training for Mentors of K-Series Mentored Career Development Awards will uniquely study mentor training in the biomedical academic community. The randomized controlled trial will be conducted at 15 Clinical and Translational Science Award sites over a 21-month period with six months for baseline data collection, nine months for the intervention, three months for follow-up, and three months for analysis. The multi-site trial will be conducted to determine whether the resultant skills-focused, case-based, mentor training program can improve the mentoring skills of K series mentors.

DETAILED DESCRIPTION:
The trial will be conducted over a 21-month period with six months for baseline data collection, nine months for the intervention, three months for follow-up, and three months for analysis. The trial will be conducted to determine whether the resultant skills-focused, case-based, mentor training program can improve the mentoring skills of K series mentors. Our modified Wisconsin Mentoring Seminar Curriculum will consist of four 2-hour sessions administered within an 8-week period, using trained facilitators. Scholars will include all recipients of a K-Series Award at the 3 CTSA sites (e.g., K01, K08, K12, K23, K24, K99, KL2), who will be funded during the two-year cycle of this Administrative Supplement. We will randomly assign 300 K-award mentors of these scholars to a control group (n=150) or to the experimental intervention (n=150).

ELIGIBILITY:
Inclusion Criteria:

- Mentor of junior faculty, post doc or PhD student engaged in clinical or translational research Willingness to attend mentor training if assigned to intervention arm

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Improvement of Mentoring Skills (comprised of 6 key competencies). | 6 months post intervention
  Based on a summative score of the 26 items assessing global mentoring skills (section 3 of the pre/post instrument) for both mentors and mentees across both the control and intervention groups.

SECONDARY OUTCOMES:
Increased Active Mentoring of the mentee | 6 months post intervention
  Based on a summative score of items in section 2 of the pre-post instrument addressing frequency of contact between mentor and mentee and the amount of review/feedback mentees receive on their grants or manuscripts for both mentors and mentees across both the control and intervention groups

CONTACTS AND LOCATIONS:
Overall Officials: Marc K Drezner, MD, Principal Investigator — UW Madison
Locations (1):
- UW Madison, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Pfund C, House SC, Asquith P, Fleming MF, Buhr KA, Burnham EL, Eichenberger Gilmore JM, Huskins WC, McGee R, Schurr K, Shapiro ED, Spencer KC, Sorkness CA. Training mentors of clinical and translational research scholars: a randomized controlled trial. Acad Med. 2014 May;89(5):774-82. doi: 10.1097/ACM.0000000000000218. PMID 24667509